CLINICAL TRIAL: NCT00769873
Title: Effect of Anticoagulation in Reducing the Incidence of Splenic/Portal Vein Thrombosis Post-Laparoscopic Splenectomy Protocol Number: 5698
Brief Title: Anticoagulation Post Laparoscopic Splenectomy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment was slower than anticipated. Insufficient funding to expand to multi-centered trial.
Sponsor: University of Alberta (Other)
Collaborators: Edmonton Civic Employees Research Fund (Other); Sanofi (Industry)
Responsible Party: Dr. James Shapiro, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5698
Record Dates: First submitted 2008-10-08; First posted 2008-10-09 (Estimated); Last update posted 2009-06-24 (Estimated); Status verified 2009-06

CONDITIONS: Portal Vein Thrombosis; Splenic Vein Thrombosis
Keywords: anticoagulation; thrombosis; portal vein thrombosis; splenic vein thrombosis; splenectomy; randomized; laparoscopic splenectomy; lovenox
MeSH Terms: conditions — Thrombosis | interventions — Enoxaparin; Heparin, Low-Molecular-Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lovenox (Active Comparator): Patients receive Lovenox 40mg SC daily (30mg SC daily if creatinine clearance < 30) for 21 days after laparoscopic splenectomy
  Interventions: Drug: Enoxaparin
- No Lovenox (No Intervention): Patients do NOT receive Lovenox post laparoscopic splenectomy

INTERVENTIONS:
Drug: Enoxaparin — Lovenox 40mg SC daily (30mg SC daily if creatinine clearance < 30) for 21 days
  Other Names: Low molecular weight heparin
  Arms: Lovenox

SUMMARY:
Splenic/portal vein thrombosis is an alarming complication of splenectomy. Retrospective studies in the literature have shown the incidence of symptomatic splenic/portal vein thrombosis to be between 0.7% (Rattner et al., 1993) to 8% (Winslow et al., 2002). This is a single-center, prospective, randomized study in subjects undergoing laparoscopic splenectomy. All participants will receive one dose of pre-operative low molecular weight heparin (Lovenox®) subcutaneously, 2 hours prior to surgery. Participants will be randomized pre-operatively to treatment or control group however the treatment allocation will not be revealed until the surgery is complete. Postoperatively, those assigned to the treatment group will receive 40 mg of Lovenox® subcutaneously once a day for 21 days; those in the control group will not. Patients with severe renal impairment will receive an adjusted dose of Lovenox® (30 mg subcutaneous dose daily). All patients will have a baseline abdominal Doppler ultrasound preoperatively and a second one done at 14 to 28 days post surgery to monitor for the presence of portal vein and/or splenic vein thrombosis. They will also have their lipase and liver function tests checked to correlate with the imaging findings.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo laparoscopic splenectomy at The University of Alberta or Grey Nun's Community Hospitals
* Capable of understanding the purpose and risks of the study and willing/able to sign a statement of informed consent
* Willing to undergo daily subcutaneous injections of Lovenox®

Exclusion Criteria:

* Pregnant or nursing
* Unable or unwilling to provide informed consent
* Bleeding diathesis or currently on anticoagulation therapy (i.e. coumadin, heparin, LMWH)
* Hemorrhagic cerebral vascular accident
* Severe uncontrolled hypertension
* Diabetic or hemorrhagic retinopathy
* Contradictions to anticoagulation (i.e. active GI bleed, gastric or duodenal ulcer, sustained platelet count < 50 x103/uL, splenectomy due to trauma or history of heparin induced thrombocytopenia)
* Conversion to open splenectomy
* Allergy to Lovenox®, heparin, or other low molecular weight heparins
* Bacterial endocarditis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2006-10; Primary Completion 2009-04 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
The incidence of portal/splenic vein thrombosis post laparoscopic splenectomy | three years

CONTACTS AND LOCATIONS:
Overall Officials: James Shapiro, MD PhD FRCS(Eng), Principal Investigator — University of Alberta; Haili Wang, MD FRCSC, Study Director — University of Alberta; Daniel Kopac, MD MSc, Study Director — University of Alberta
Locations (2):
- Canada (2):
  - University of Alberta Hospital, Edmonton, Alberta
  - Grey Nuns Hospital, Edmonton, Alberta

REFERENCES:
- [Background] Bergqvist D, Agnelli G, Cohen AT, Eldor A, Nilsson PE, Le Moigne-Amrani A, Dietrich-Neto F; ENOXACAN II Investigators. Duration of prophylaxis against venous thromboembolism with enoxaparin after surgery for cancer. N Engl J Med. 2002 Mar 28;346(13):975-80. doi: 10.1056/NEJMoa012385. PMID 11919306
- [Background] Bergqvist D. Low molecular weight heparin for the prevention of venous thromboembolism after abdominal surgery. Br J Surg. 2004 Aug;91(8):965-74. doi: 10.1002/bjs.4639. PMID 15286956
- [Background] Chaffanjon PC, Brichon PY, Ranchoup Y, Gressin R, Sotto JJ. Portal vein thrombosis following splenectomy for hematologic disease: prospective study with Doppler color flow imaging. World J Surg. 1998 Oct;22(10):1082-6. doi: 10.1007/s002689900521. PMID 9747171
- [Background] Efficacy and safety of enoxaparin versus unfractionated heparin for prevention of deep vein thrombosis in elective cancer surgery: a double-blind randomized multicentre trial with venographic assessment. ENOXACAN Study Group. Br J Surg. 1997 Aug;84(8):1099-103. PMID 9278651
- [Background] Fujita F, Lyass S, Otsuka K, Giordano L, Rosenbaum DL, Khalili TM, Phillips EH. Portal vein thrombosis following splenectomy: identification of risk factors. Am Surg. 2003 Nov;69(11):951-6. PMID 14627254
- [Background] Geerts WH, Pineo GF, Heit JA, Bergqvist D, Lassen MR, Colwell CW, Ray JG. Prevention of venous thromboembolism: the Seventh ACCP Conference on Antithrombotic and Thrombolytic Therapy. Chest. 2004 Sep;126(3 Suppl):338S-400S. doi: 10.1378/chest.126.3_suppl.338S. PMID 15383478
- [Background] Mismetti P, Laporte S, Darmon JY, Buchmuller A, Decousus H. Meta-analysis of low molecular weight heparin in the prevention of venous thromboembolism in general surgery. Br J Surg. 2001 Jul;88(7):913-30. doi: 10.1046/j.0007-1323.2001.01800.x. PMID 11442521
- [Background] Petit P, Bret PM, Atri M, Hreno A, Casola G, Gianfelice D. Splenic vein thrombosis after splenectomy: frequency and role of imaging. Radiology. 1994 Jan;190(1):65-8. doi: 10.1148/radiology.190.1.8259430.
- [Background] van't Riet M, Burger JW, van Muiswinkel JM, Kazemier G, Schipperus MR, Bonjer HJ. Diagnosis and treatment of portal vein thrombosis following splenectomy. Br J Surg. 2000 Sep;87(9):1229-33. doi: 10.1046/j.1365-2168.2000.01514.x. PMID 10971433